CLINICAL TRIAL: NCT06941883
Title: A Study of Ultrasound-Guided Versus Anatomically Guided Botulinum Toxin Injection in Spasticity in Adults in Tanta University Hospitals
Brief Title: Ultrasound-Guided Versus Anatomically Guided Botulinum Toxin Injection in Spasticity in Adults in Tanta University Hospitals
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Omar Abdallah Ebrahim Elsaharty, Resident of Neuropsychiatry, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264MS248/7/23
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ultrasound; Botulinum Toxin; Spasticity; Adults
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Botulinum toxin injection under anatomical landmark: Patients received botulinum toxin injections under the anatomical landmark.
  Interventions: Drug: Botulinum toxin injection under anatomical landmark
- Ultrasound-guided botulinum toxin injection: Patients received ultrasound-guided botulinum toxin injection
  Interventions: Drug: Ultrasound-guided botulinum toxin injection

INTERVENTIONS:
Drug: Botulinum toxin injection under anatomical landmark — Patients received botulinum toxin injections under the anatomical landmark.
  Groups: Botulinum toxin injection under anatomical landmark
Drug: Ultrasound-guided botulinum toxin injection — Patients received ultrasound-guided botulinum toxin injection
  Groups: Ultrasound-guided botulinum toxin injection

SUMMARY:
This study aimed to compare the safety and outcome of ultrasound (US)- guided botulinum toxin (BoNT) injection and anatomically guided injection in muscle spasticity of different causes in adults.

DETAILED DESCRIPTION:
One of the major complications of neurological diseases is spasticity which is defined as an increased velocity-dependent muscle tone.

A large volume of clinical data has demonstrated the efficacy and safety of botulinum toxin type A (BoNT-A) products for treating conditions such as spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Both sexes.
* Patients with muscle spasticity.

Exclusion Criteria:

- Patients with contraindications to botulinum toxin injection as allergy, myasthenia gravis, and cerebral palsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective case-controlled study was carried out on 68 patients aged > 18 years old, both sexes, with muscle spasticity, planned and indicated for BoNT injection according to recent guidelines. The study was done from July 2023 to July 2024 after approval from the Ethical Committee Tanta University Hospitals, Tanta, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment the range of movement | 6 months after the procedure
  The range of movement regarding forearm pronation, thumb flexion, ankle inversion and fingers flexion according to modified Ashworth scale (MAS): score zero indicate no increase in tone, score 1 indicate slight increase in tone, catch or release at end range of motion (ROM), score 1 + indicate a slight increase in tone catch, release, resistance through rest ROM (1/2 ROM), score 2 indicate more marked increase in tone through ROM but affected part moved easily, score 3 indicate a considerable increase in tone, passive movement difficult, score 4 indicate affected part in rigid flexion and extension. It was assessed after three and six months.

SECONDARY OUTCOMES:
Assessment the quality of life | 6 months after the procedure
  Patients' quality of life (QOL) was assessed before and after intervention with the World Health Organization (WHO)-QOL scale). The WHOQOL is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.